CLINICAL TRIAL: NCT04970251
Title: Aflibercept as Adjunctive Treatment for Filtration Surgery in Neovascular
Brief Title: Aflibercept as Adjunctive Treatment for Filtration Surgery in Neovascular Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Naris Kitnarong, Associate professor, Siriraj Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Si726/2018
Record Dates: First submitted 2021-06-24; First posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Intraocular Pressure; Neovascular Glaucoma; Vascular Endothelial Growth Factor Overexpression; Glaucoma Secondary to Eye Inflammation
MeSH Terms: conditions — Glaucoma, Neovascular | interventions — Trabeculectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Aflibercept Ophthalmic — Panretinal photocoagulation and intravitreal aflibercept (2 mg/0.05 ml) injection were given, and trabeculectomy with mitomycin C was performed within 2 weeks after intravitreal aflibercept injection.
  Other Names: trabeculectomy; Panretinal photocoagulation

SUMMARY:
Purpose: To investigate intravitreal aflibercept (IVA) injection as an adjunctive treatment to trabeculectomy with mitomycin C (TMC) and panretinal photocoagulation (PRP) for neovascular glaucoma (NVG).

Setting: Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Thailand Study design: Prospective interventional case series Methods: PRP and IVA (2 mg/0.05 ml) injection were given, and TMC was performed within 2 weeks after IVA. Additional PRP, laser suture lysis, subconjunctival 5-fluorouracil injection, and bleb needling were performed after TMC if indicated. Best-collected visual acuity (BCVA), intraocular pressure (IOP), surgical complications, and number of anti-glaucoma medications were collected.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with neovascular glaucoma who presented at the Department of Ophthalmology, Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Thailand during November 2018 to October 2019.
* Aged more than 18 year-old

Exclusion Criteria:

* Patients who received any anti-vascular endothelial growth factor treatment before participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure | Post-operative on day 1st
  Intraocular pressure after trabeculectomy
Intraocular pressure | Post-operative on day 7th
  Intraocular pressure after trabeculectomy
Intraocular pressure | Post-operative on month 3rd
  Intraocular pressure after trabeculectomy
Intraocular pressure | Post-operative on month 6th
  Intraocular pressure after trabeculectomy
Intraocular pressure | Post-operative on month 12th
  Intraocular pressure after trabeculectomy
Intraocular pressure | Post-operative on month 18th
  Intraocular pressure after trabeculectomy
Intraocular pressure | Post-operative on month 24th
  Intraocular pressure after trabeculectomy
Intraocular pressure | Post-operative on month 30th
  Intraocular pressure after trabeculectomy
Intraocular pressure | Post-operative on month 36th
  Intraocular pressure after trabeculectomy

SECONDARY OUTCOMES:
Visual acuity | Post-operative on day 1st
  Visual acuity of the studied eye
Visual acuity | Post-operative on day 7th
  Visual acuity of the studied eye
Visual acuity | Post-operative on month 3rd
  Visual acuity of the studied eye
Visual acuity | Post-operative on month 6th
  Visual acuity of the studied eye
Visual acuity | Post-operative on month 12th
  Visual acuity of the studied eye
Visual acuity | Post-operative on month 18th
  Visual acuity of the studied eye
Visual acuity | Post-operative on month 24th
  Visual acuity of the studied eye
Visual acuity | Post-operative on month 30th
  Visual acuity of the studied eye
Visual acuity | Post-operative on month 36th
  Visual acuity of the studied eye
Numbers of medication | Post-operative on month12th
  Numbers of anti-glaucoma medications
Numbers of medication | Post-operative on month 24th
  Numbers of anti-glaucoma medications
Numbers of medication | Post-operative on month 36th
  Numbers of anti-glaucoma medications

CONTACTS AND LOCATIONS:
Locations (1):
- Naris Kitnarong, Bangkoknoi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided
Centers who collect the data of neovascular Glaucoma patients who underwent intravitreal aflibercept injection, pan retinal photocoagulation and trabeculectomy with mitomycin C.

REFERENCES:
- [Result] Kitnarong N, Sriyakul C, Chinwattanakul S. A Prospective Study to Evaluate Intravitreous Ranibizumab as Adjunctive Treatment for Trabeculectomy in Neovascular Glaucoma. Ophthalmol Ther. 2015 Jun;4(1):33-41. doi: 10.1007/s40123-015-0033-3. Epub 2015 Mar 27. PMID 25812531
- [Result] Kitnarong N, Chindasub P, Metheetrairut A. Surgical outcome of intravitreal bevacizumab and filtration surgery in neovascular glaucoma. Adv Ther. 2008 May;25(5):438-43. doi: 10.1007/s12325-008-0047-5. PMID 18425438
- [Result] Kobayashi S, Inoue M, Yamane S, Sakamaki K, Arakawa A, Kadonosono K. Long-term Outcomes After Preoperative Intravitreal Injection of Bevacizumab Before Trabeculectomy for Neovascular Glaucoma. J Glaucoma. 2016 Mar;25(3):281-4. doi: 10.1097/IJG.0000000000000211. PMID 25580888